CLINICAL TRIAL: NCT01396928
Title: Prospective Randomized Study of Two Techniques of Rectal Reservoir in Low Anterior Resection of Rectum
Brief Title: Study of Two Techniques of Rectal Reservoir in Low Anterior Resection of Rectum
Status: Completed | Type: Observational
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Sebastiano Biondo, MD, Barcelona University
Other Study IDs: CGD-01/2000
Record Dates: First submitted 2011-07-18; First posted 2011-07-19 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2000-11

CONDITIONS: Low Rectal Adenocarcinoma
Keywords: Low rectal adenocarcinoma
MeSH Terms: interventions — Urinary Reservoirs, Continent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- "J" pouch: Anastomosis coloanal wiht "j" pouch reservoir
  Interventions: Procedure: Colonic reservoir
- Transverse coloplasty pouch: Coloanal anastomosis with transverse coloplasty pouch reservoir
  Interventions: Procedure: Colonic reservoir

INTERVENTIONS:
Procedure: Colonic reservoir — Type of reservoir to be performed

SUMMARY:
The aim of the study CGD-01/2000 was to investigate wheter a transverse coloplasty pouch is able to improve functional results and quality of life after coloanal anastomosis.

ELIGIBILITY:
Inclusion Criteria:

* Low or middle rectal adenocarcinoma without involvement of the anal sphincter
* Neoadjuvant chemoradiotherapy
* Age older than 18 years
* Wexner index of less than 5
* Signed informed consent

Exclusion Criteria:

* Involvement of the anal sphincter
* Wexner index of 5 or more
* Declined informed consent
* Psychological or social problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients wiht low or middle rectal adenocarcinoma after neoadyuvant radio-chemotherapy
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2000-11; Primary Completion 2005-12 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Quality of life | five years
  Functional results and quality of life after coloanal anastomosis with colonic reservoir

SECONDARY OUTCOMES:
Morbidity and cost-effectiveness | 30 days
  Investigate if the new technique is more easily, quickly and cheap.

REFERENCES:
- [Derived] Biondo S, Frago R, Codina Cazador A, Farres R, Olivet F, Golda T, Miguel B, Kreisler E. Long-term functional results from a randomized clinical study of transverse coloplasty compared with colon J-pouch after low anterior resection for rectal cancer. Surgery. 2013 Mar;153(3):383-92. doi: 10.1016/j.surg.2012.08.012. Epub 2012 Sep 14. PMID 22981362